CLINICAL TRIAL: NCT06727656
Title: Exercise in Hypoxia and Nitrate Supplementation in Athletes: is the Whole Greater Than the Sum of Its Parts?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Responsible Party: Principal Investigator, Ana Sousa, PhD, Advanced Bionics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hypoxia
Record Dates: First submitted 2024-07-24; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HNO: High intensity interval training (HIIT) + nitrate supllementation (NO3-). (Experimental): Performed 12 high-intensity interval-training (HIIT) sessions during a 4-week period (3 sessions/ week) under normobaric hypoxia conditions (FiO2=~13%, ~3000 m) with NO3- supplement.
  Interventions: Combination Product: Nitrate + Hypoxia
- HPL: High intensity interval training (HIIT) + placebo supllementation. (Active Comparator): Performed 12 high-intensity interval-training (HIIT) sessions during a 4-week period (3 sessions/ week) under normobaric hypoxia conditions (FiO2=~13%, ~3000 m) with placebo supplement.
  Interventions: Dietary Supplement: Placebo + Hypoxia
- CON: High intensity interval training (HIIT) + placebo supllementation. (Placebo Comparator): Performed 12 high-intensity interval-training (HIIT) sessions during a 4-week period (3 sessions/ week) under normoxic conditions (FiO2=~20.9%) with placebo supplement.
  Interventions: Other: Control

INTERVENTIONS:
Combination Product: Nitrate + Hypoxia — The combined effect of nitrate supplementation and hypoxia training on both performance and health at sea-level and altitude conditions.
  Other Names: Beetroot Juice + Atitude training
  Arms: HNO: High intensity interval training (HIIT) + nitrate supllementation (NO3-).
Dietary Supplement: Placebo + Hypoxia — The combined effect of placebo supplementation and hypoxia training on both performance and health at sea-level and altitude conditions.
  Other Names: Placebo Juice + Atitude training
  Arms: HPL: High intensity interval training (HIIT) + placebo supllementation.
Other: Control — The combined effect of placebo supplementation and normoxia training on both performance and health at sea-level and altitude conditions.
  Other Names: Placebo Juice + Normoxia training
  Arms: CON: High intensity interval training (HIIT) + placebo supllementation.

SUMMARY:
Determine the combined effect of training in hypoxia and nitrate supplementation on the performance and health of athletes at sea-level and altitude conditions.

DETAILED DESCRIPTION:
Determine the combined effect of training in hypoxia and nitrate supplementation on the performance and health of athletes at sea-level and altitude conditions. It is hypothesized that the combined effect of these interventions will promote an additional performance and health improvement in this population at sea-level and altitude conditions, compared with the single effect.

ELIGIBILITY:
Inclusion Criteria:

* trained male subjects, regularly involved in competitive running, cycling and/ or triathlon events (4-5 times per week) in the past five years

Exclusion Criteria:

* smoking or other chronic issues
* using medication or dietary supplements in the last 3 months, or during the duration of the study
* being exposed to altitude (≥2000 m) in the last 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Performance adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Time-to-task failure (time sustained)
Performance adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Time trials (time performed)
Performance adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  VO2 kinetics (time constant and amplitude of fast and slow oxygen components)
Cardiovascular and neuromuscular adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Maximal oxygen uptake (VO2max: absolute and relative value)
Cardiovascular and neuromuscular adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Lactate threshold (absolute and percentage of VO2max)
Cardiovascular and neuromuscular adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Muscular oxygen saturation (SmO2)
Skeletal muscle adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Oxidative enzyme activity (cytochrome oxidase subunit IV), citrate synthase, transcription factors (HIF-1alpha and PGC-1alpha) and GLUT4 - assessed through standard enzymatic fluorometric assay and western bllotting
Skeletal muscle adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Mitochondrial and capillary density, capillary-to-fibre ratio and fibre cross-section area - cryosections cut with a cryostat and further samples analysed by fluorescence microscopy
Haematological adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Blood pressure (Hmmg), mean arterial pressure (calculated as 1/3 * systolic pressure + 2/3 * diastolic pressure)
Haematological adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Plasma [NO2-] and [NO3-], erythropoietin (EPO), haemoglobin (Hb) and haematocrit (Hct) - all assays on plasma sample analysed by spectrophometry
Oxidative stress and antioxidant markers adaptations | Moment #1 (48hours pre-intervention) and moment #2 (48hours post-intervention)
  Nitrotyrosine, malondialdehyde, ferric-reducing antioxidant power and superoxide dismutase concentrations - all assays on plasma sample analysed by spectrophometry

SECONDARY OUTCOMES:
Sleep and cardiac autonomic activity adaptations | Moment #1 (2 weeks pre-intervention - baseline) and moment #2 (4 weeks intervention)
  Sleep duration (minutes)
Sleep and cardiac autonomic activity adaptations | Moment #1 (2 weeks pre-intervention - baseline) and moment #2 (4 weeks intervention)
  Sleep efficiency (%)
Sleep and cardiac autonomic activity adaptations | Moment #1 (2 weeks pre-intervention - baseline) and moment #2 (4 weeks intervention)
  Wake up time (hours: minutes)
Sleep and cardiac autonomic activity adaptations | Moment #1 (2 weeks pre-intervention - baseline) and moment #2 (4 weeks intervention)
  Resting heart rate (bpm)
Sleep and cardiac autonomic activity adaptations | Moment #1 (2 weeks pre-intervention - baseline) and moment #2 (4 weeks intervention)
  Heart rate variability (lnRMSSD)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Sousa, PhD, Principal Investigator — University of Maia
Locations (1):
- University of Trás-os-Montes e Alto-Douro, Vila Real, Portugal

IPD SHARING:
Plan to Share IPD: No
Study overview, participation criteria, study plan, contacts